CLINICAL TRIAL: NCT03353688
Title: Noninvasive Biomarkers to Advance Emerging DBS Electrode Technologies in Parkinson's Disease (SUNDIAL, SUbthalamic Nucleus DIrectionAL vs Circular Stimulation Study)
Brief Title: Biomarkers to Guide Directional DBS for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Harrison Walker, MD, Professor of Neurology, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-161018001; 1UH3NS100553-01 (NIH)
Record Dates: First submitted 2017-09-26; First posted 2017-11-27 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a triple blind, randomized crossover study of directional versus omnidirectional unilateral subthalamic deep brain stimulation for Parkinson's disease with motor fluctuations.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a triple blind study. Participants, raters, and investigator are masked to the assignment of directional versus omnidirectional unilateral subthalamic deep brain stimulation guided by behavioral programming for Parkinson's disease with motor fluctuations. For the nested exploratory arm evaluating directional DBS guided by electrophysiology biomarkers, the study is double-blind (investigator is not blinded).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Directional DBS guided by behavior (Active Comparator): Directional stimulation with the Boston Scientific Vercise PC IPG with directional DBS lead, guided by behavioral assessments during device activation.
  Interventions: Device: Boston Scientific Vercise PC IPG with directional DBS lead
- Omnidirectional DBS guided by behavior (Placebo Comparator): Omnidirectional ("ring mode") stimulation with the Boston Scientific Vercise PC IPG with directional DBS lead, guided by behavioral assessments during device activation.
  Interventions: Device: Boston Scientific Vercise PC IPG with directional DBS lead
- Directional DBS guided by biomarkers (Active Comparator): Directional unilateral subthalamic stimulation with the Boston Scientific Vercise PC IPG with directional DBS lead, guided by electrophysiology biomarkers measured during surgery (nested exploratory treatment arm).
  Interventions: Device: Boston Scientific Vercise PC IPG with directional DBS lead

INTERVENTIONS:
Device: Boston Scientific Vercise PC IPG with directional DBS lead — Deep brain stimulation

SUMMARY:
The purpose of this study is to investigate the clinical efficacy of directional DBS electrode technology and whether electrophysiology biomarkers can predict effective contact segments for chronic therapy.

DETAILED DESCRIPTION:
Although deep brain stimulation (DBS) can be remarkable for treating symptoms of Parkinson's disease, improvement varies across clinical trials, individual patients, and over time. A major limitation to the advancement of DBS therapy is that there are no established biomarkers to tailor stimulator settings in individuals. Emerging segmented ("directional") lead technology allows current steering, a new opportunity to improve tolerability and efficacy by shaping the DBS electrical field. This novel lead design has 8 contacts rather than the 4 available with currently available leads. How do the investigators optimally adjust stimulation parameters when there are far more potentially useful settings than can be practically evaluated in clinic? How do the investigators know that DBS settings in a given patient are optimal or appropriate? The investigators have pioneered minimally invasive, rapidly acquired biomarkers to solve these important problems. Using electrocorticography, electroencephalography, and subcortical local field potentials, the investigators will measure whether resting or stimulus-evoked electrophysiology can serve as a predictive biomarker to guide activation and adjustment of a directional DBS system. The purpose of this randomized, double-blind crossover study is to measure the clinical efficacy of directional versus omnidirectional stimulation and to explore whether electrophysiology biomarkers can rapidly predict effective, well-tolerated contacts for directional DBS therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤70 years.
2. Clinically definite, advanced idiopathic PD based on at least 2 of 3 cardinal PD features (tremor, rigidity, or bradykinesia).
3. Disease duration of 4 years or more.
4. Participant has elected to undergo DBS surgery as part of routine care, and the subthalamic nucleus (STN) is recommended as the surgical target.
5. Participant agrees to not undergo contralateral DBS for the other side of the brain until ≥ 12 months after initial DBS surgery.
6. Participant is healthy enough to undergo surgery and the research protocol.
7. Normal, or essentially normal, preoperative brain MRI.
8. Willingness and ability to cooperate during awake DBS surgery, as well as during post-operative evaluations, adjustments of medications and stimulator settings.
9. Participant's health insurance and/or Medicare covers DBS surgery as part of routine care.
10. Refractory motor symptoms such as tremor, dyskinesias, wearing off, and/or motor fluctuations, causing significant disability or occupational dysfunction, despite reasonable attempts at medical management, as determined by our consensus DBS committee.
11. Stable doses of PD medications for at least 28 days prior to baseline assessments.
12. Improvement of motor signs ≥30% with dopaminergic medication as assessed with the use of the Movement Disorders - Unified Parkinson's Disease Rating Scale, part III (MDS-UPDRS III; scores range from 0 to 108, with higher scores indicating worse functioning).
13. Disease severity ratings above Hoehn and Yahr stage 1, defined as unilateral involvement only with minimal or no functional disability, with scores ranging from 0 to 5 and higher scores indicating more severe disease.
14. Score of more than 6 for activities of daily living in the worst "off" medication condition despite medical treatment, as assessed with the use of the MDS-UPDRS II (scores range from 0 to 52, with higher scores indicating worse functioning), or mild-to-moderate impairment in social and occupational functioning (score of 51 to 80% on the Social and Occupational Functioning Assessment Scale with scores ranging from 1 to 100 and lower scores indicating worse functioning).
15. Dementia Rating Scale-2 (DRS-2) score of ≥130 on medications.
16. Beck Depression Inventory II (BDI-II) score of ≤25 on medications.
17. Participant expresses understanding of the consent process, terms of the study protocol, is available for follow-up over the length of the study, and signs informed consent.

Exclusion Criteria:

1. Age <18 years or >70 years.
2. Participant's insurance will not cover the costs of surgery with the investigational device.
3. Medical contraindications such as current uncontrolled hypertension, heart disease, coagulopathy, or other conditions contraindicating DBS surgery or stimulation.
4. Duration of disease of <4 years
5. Participant or care team determine that contralateral DBS for the other side of the brain will likely be clinically indicated <12 months after initial DBS surgery.
6. Diagnosis or suspicion of atypical parkinsonism (progressive supranuclear palsy, multiple system atrophy, corticobasal syndrome) or drug-induced parkinsonism, or significant neurological disease other than Parkinson's disease.
7. Disease severity ratings of Hoehn and Yahr stage 1, defined as unilateral involvement only with minimal or no functional disability, with scores ranging from 0 to 5 and higher scores indicating more severe disease.
8. Diagnosis of psychogenic movement disorder based on consensus criteria.
9. Score of >25 on the Beck Depression Inventory II, with scores ranging from 0 to 63 and higher scores indicating worse functioning), or history of suicide attempt.
10. Any current acute psychosis, alcohol abuse or drug abuse.
11. Clinical dementia (score of ≤130 on the Mattis Dementia Rating Scale with scores ranging from 0 to 144 and higher scores indicating better functioning).
12. Ongoing or pervasive impulse control disorder not resolved by reduction of dopaminergic medications.
13. Use of anticoagulant medications that cannot be discontinued during perioperative period.
14. History of hemorrhagic stroke.
15. Current or future risk of immunocompromise that might significantly increase risk of infection.
16. History of recurrent of unprovoked seizures.
17. Lack of clear levodopa responsiveness.
18. Any medical condition requiring repeated MRI.
19. The presence of an implanted device (e.g., cochlear implant, pacemaker, neurostimulators), whether turned on or off.
20. Prior DBS surgery or ablation within the affected basal ganglion.
21. A condition requiring or likely to require the use of diathermy.
22. Structural lesions such as basal ganglionic stroke, tumor or vascular malformation as etiology of the movement disorder.
23. Any medical or psychological problem that would interfere with the conduction of the study protocol
24. A female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Walker, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share data through the Data Archive BRAIN Initiative (DABI) data sharing consortium.
Supporting Information: CSR, Analytic Code
Time Frame: The data will be made available after analyses of the primary and secondary outcomes.
Access Criteria: Users must set up an account on the DABI website to be able to access data.
URL: https://dabi.loni.usc.edu/

REFERENCES:
- [Derived] Black SD, Del Bene VA, Celka AS, Guthrie B, Martin RC, Olson J, Shumake J, Walker HC. Nascent visual artistic expression following right hemisphere subthalamic nucleus deep brain stimulation for Parkinson's disease. Parkinsonism Relat Disord. 2022 Jun;99:47-50. doi: 10.1016/j.parkreldis.2022.04.020. Epub 2022 May 1. No abstract available. PMID 35598419

RESULTS

PARTICIPANT FLOW:
Groups:
- Directional DBS by Behavior; Omnidirectional DBS by Behavior; Directional DBS by Biomarkers Last: Participants were randomly assigned to directional stimulation with the Boston Scientific Vercise PC IPG with directional DBS lead, guided by behavioral assessments. Next they were assigned to omnidirectional stimulation based on behavior. Finally, they were assigned to directional DBS based on biomarkers recorded in surgery.
  First Intervention (2 months), Second Intervention (2 months), and Third Intervention (2 months).
- Omnidirectional DBS by Behavior; Directional DBS by Behavior; Directional DBS by Biomarkers Last: Participants were randomly assigned to omnidirectional stimulation with the Boston Scientific Vercise PC IPG with directional DBS lead, guided by behavioral assessments. Next they were assigned to directional stimulation based on behavior. Finally, they were assigned to directional DBS based on biomarkers recorded in surgery.
  First Intervention (2 months), Second Intervention (2 months), and Third Intervention (2 months).
- Either Directional DBS or Omnidirectional DBS by Behavior; Directional DBS by Biomarkers Last: Upon completion of the first two periods (either directional stimulation or omnidirectional stimulation based on behavioral assessments), all participants were assigned to a directional unilateral subthalamic stimulation strategy with the Boston Scientific Vercise PC IPG with directional DBS lead, guided by electrophysiology biomarkers measured during surgery (nested exploratory treatment arm).
  First Intervention (2 months), Second Intervention (2 months), and Third Intervention (2 months).
Period: First Intervention (2 Months)
Arm/Group | Directional DBS by Behavior; Omnidirectional DBS by Behavior; Directional DBS by Biomarkers Last | Omnidirectional DBS by Behavior; Directional DBS by Behavior; Directional DBS by Biomarkers Last | Either Directional DBS or Omnidirectional DBS by Behavior; Directional DBS by Biomarkers Last
Started | 17 | 14 | 0
Completed | 17 | 14 | 0
Not Completed | 0 | 0 | 0
Period: Second Intervention (2 Months)
Arm/Group | Directional DBS by Behavior; Omnidirectional DBS by Behavior; Directional DBS by Biomarkers Last | Omnidirectional DBS by Behavior; Directional DBS by Behavior; Directional DBS by Biomarkers Last | Either Directional DBS or Omnidirectional DBS by Behavior; Directional DBS by Biomarkers Last
Started | 14 | 17 | 0
Completed | 14 | 17 | 0
Not Completed | 0 | 0 | 0
Period: Third Intervention (2 Months)
Arm/Group | Directional DBS by Behavior; Omnidirectional DBS by Behavior; Directional DBS by Biomarkers Last | Omnidirectional DBS by Behavior; Directional DBS by Behavior; Directional DBS by Biomarkers Last | Either Directional DBS or Omnidirectional DBS by Behavior; Directional DBS by Biomarkers Last
Started | 0 | 0 | 31
Completed | 0 | 0 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 31 participants experienced all arms of the study.
Groups:
- All Study Participants: Aggregate baseline data for all study participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.85 (7.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Preoperative Baseline in Movement Disorders Society Unified Parkinson's Disease Rating Scale Part 3 (MDS-UPDRS Part III) "Off" Medications
Description: A blinded examiner will measure Movement Disorders Society Unified Parkinson's Disease Rating Scale Part 3 motor scores "off" medications. MDS-UPDRS Part III is a motor examination consisting of 18 summed items where the investigator rates the severity of Parkinson's motor symptoms based on a scale of 0 - 4. Higher values indicate worse function (possible min score = 0, possible max score = 72).
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -16.90322581 (9.253305135) | -15.80645161 (9.257139064) | -18.33333333 (9.848274252)

2. Primary Outcome: Treatment Preference Survey Programming Strategy Preference
Description: Based on overall quality of life, participants will select their preference between directional and omnidirectional DBS.
Time Frame: 4 months post surgery
Population: All participants experienced all three arms of the crossover study.
Measure: Count of Participants; unit: Participants
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior
Number analyzed (Participants) | 30 | 30
Participants | 16 | 14

3. Secondary Outcome: Change From Preoperative Baseline in the Beck Depression Inventory-2 (BDI-2)
Description: The Beck Depression Inventory-2 is a 21 question self-report inventory which evaluates a person's severity of depression. Items are answered on a 0 - 3 scale. Higher values indicate worse function (possible min score = 0, possible max score = 63).
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 0.965517241 (6.455798936) | 1.032258065 (5.056242814) | 0.692307692 (6.739550316)

4. Secondary Outcome: Change From Preoperative Baseline in the Beck Anxiety Inventory (BAI)
Description: The Beck Anxiety Inventory is a 21 question self-report inventory which evaluates a person's severity of anxiety. Items are answered on a 0 - 3 scale. Higher values indicate worse function (possible min score = 0, possible max score = 63).
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -2.55 (5.689093906) | -0.333333333 (6.32455532) | -0.6875 (8.16266909)

5. Secondary Outcome: Change From Preoperative Baseline in the Auditory Verbal Learning Test (AVLT) Delayed Recall Raw Score (Versions AB, CD, CR, GE)
Description: The Auditory Verbal Learning Test (AVLT) delayed recall raw score (versions AB, CD, CR, GE) evaluates a person's ability to encode, consolidate, store, and retrieve verbal information. Participants are read a list of 12 words and later asked to recall the items on the list. Scores indicate the number of items recalled. Higher values indicate better function (possible min score = 0, possible max score = 12).
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -0.866666667 (3.785027976) | -0.9 (3.39726056) | -0.461538462 (3.776037809)

6. Secondary Outcome: Change From Preoperative Baseline in the Auditory Verbal Learning Test (AVLT) Recognition Raw Score (Versions AB, CD, CR, GE)
Description: The Auditory Verbal Learning Test (AVLT) Recognition Raw Score (versions AB, CD, CR, GE) evaluates a person's ability to encode, consolidate, store, and retrieve verbal information. Participants are given a list of 15 target words. The list is taken away and each is asked to now pick out the 15 target words from a larger list of 30 words. Scores indicate the overall number of target words correctly recognized (minimum = 0, maximum = 15). Higher scores indicate better performance.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -0.5 (1.696853071) | -0.433333333 (1.59056124) | -0.961538462 (1.482720991)

7. Secondary Outcome: Change From Preoperative Baseline in the Auditory Verbal Learning Test (AVLT) Learning Raw Score (Versions AB, CD, CR, GE)
Description: The AVLT (versions AB, CD, CR, GE) evaluates a person's ability to encode, consolidate, store, and retrieve verbal information. Participants are read a list of 12 words and asked to immediately recall the items on the list over 6 separate trials. Scores indicate the number of items recalled. Higher values indicate better function (possible min score = 0, possible max score = 72).
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -2.233333333 (9.772174901) | -3.3 (9.203260292) | -0.576923077 (8.276100903)

8. Secondary Outcome: Change From Preoperative Baseline in the Letter Fluency Test Raw Score (Version: CFL, FAS)
Description: The Letter Fluency Test (version: CFL, FAS) evaluates the number of words beginning with the letters C, F, L, A, and S that a participant can produce in one minute (minimum = 0, maximum = infinity). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: words generated
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
words generated | -1.766666667 (8.21975473) | -1.935483871 (9.401898687) | -1.230769231 (9.074393389)

9. Secondary Outcome: Change From Preoperative Baseline in the Voice Handicap Index
Description: The Voice Handicap Index evaluates speech function with a 30-item self-administered questionnaire that asks participants to describe their voice and the effects of their voice on their lives. Participants respond on a 0 - 4 scale (minimum = 0, maximum = 120. Higher scores indicate worse functiion.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -2.709677419 (9.256325939) | 0.225806452 (7.774786931) | -0.925925926 (12.04135798)

10. Secondary Outcome: Change From Preoperative Baseline in the Communicative Participation Item Bank (CPIB)
Description: The Communicative Participation Item Bank (CPIB) evaluates the extent to which communication disorders interfere with communicative participation. Participants respond on a 0 - 3 scale (minimum = 0, maximum = 30). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -0.387096774 (3.489769996) | -0.741935484 (2.920818857) | -0.740740741 (4.927103944)

11. Secondary Outcome: Change From Preoperative Baseline in the 9-Hole Pegboard Test
Description: The 9-Hole Pegboard Test evaluates one's upper extremity motor function. It is a timed test in which participants place 9 pegs in a pegboard and then remove them. Faster times indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: time (seconds)
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
time (seconds) | -6.15 (10.86369404) | -5.242258065 (11.16955019) | -6.755 (11.38578962)

12. Secondary Outcome: Change From Preoperative Baseline in Gait Initiation Test
Description: The gait initiation test evaluates the phase between standing motionless and steady-state locomotion. This is a timed test in which participants are given a go signal and the time until first stride is recorded. Faster times indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: time (seconds)
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
time (seconds) | 5.810333333 (22.17604991) | 2.491 (22.48954996) | 2.282 (27.67356219)

13. Secondary Outcome: Change From Preoperative Baseline in Stepping Thresholds Test
Description: The stepping thresholds test evaluates a person's compensatory stepping thresholds. This is a test in which the floor surface is unexpectedly moved beneath a participant. The distance a participant moves their feet in order to compensate is recorded. The smaller displacement scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: mm displacement
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
mm displacement | 0.616666667 (0.762067665) | 0.583333333 (0.732065257) | 0.603448276 (0.76039593)

14. Secondary Outcome: Change From Preoperative Baseline in Quiet Stance Measure
Description: The quiet stance measure evaluates a person's postural control during quiet standing. This is a measure of sway distance. Lower scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline mm sway
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline mm sway | -243.7980645 (746.4082743) | -50.747 (819.179683) | -65.52133333 (966.9356483)

15. Secondary Outcome: Change From Preoperative Baseline in the Parkinson's Disease Quality of Life
Description: The Parkinson's Disease Quality of Life (PDQ-8) evaluates overall health status. It consists of eight questions regarding mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. Participants choose answers on a scale ranging from never (0) to always (4) (minimum = 0, maximum = 32). Higher scores indicate worse function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -5.756833333 (11.44863367) | -6.274655172 (12.96997528) | -7.924615385 (14.85058274)

16. Secondary Outcome: Change From Preoperative Baseline in the the Neuro-QOL Item Bank v1.0 "Positive Affect and Well-Being" Short Form
Description: The Neuro-QOL Item Bank v1.0 "Positive Affect and Well-Being" Short Form evaluates feelings that reflect a level of general satisfaction with life as well as a sense that life has purpose and meaning. Participants respond to questions on a 1-5 scale (minimum = 9, maximum = 45). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 1.321428571 (5.34064479) | 0.1 (5.652890625) | 0.04 (3.469870315)

17. Secondary Outcome: Change From Preoperative Baseline in the Neuro-QOL Item Bank v1.1 "Satisfaction With Social Roles and Activities" Short Form
Description: The Neuro-QOL Item Bank v1.1 "Satisfaction with Social Roles and Activities" short form short form evaluates one's satisfaction and discontentment with performing usual social roles and activities. Participants respond to questions on a 1-5 scale (minimum = 8, maximum = 40). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 2.142857143 (4.352217704) | 3.586206897 (4.917296305) | 1.24 (4.064890322)

18. Secondary Outcome: Change From Preoperative Baseline in the Neuro-QOL Item Bank v2.0 "Cognitive Function" Short Form
Description: The Neuro-QOL Item Bank v2.0 ""Cognitive Function" short form evaluates mental acuity, concentration, verbal and nonverbal memory, verbal fluency, and perceived changes in these cognitive functions. Participants respond to questions on a 1-5 scale (minimum = 8, maximum = 40). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 3.821428571 (4.83853032) | 3.333333333 (5.234720513) | 2.72 (6.045108215)

19. Secondary Outcome: Change From Preoperative Baseline in the Neuro-QOL Item Bank v1.0 "Lower Extremity Function (Mobility)" Short Form
Description: The Neuro-QOL Item Bank v1.0 "Lower Extremity Function (Mobility)" short form evaluates functioning of one's lower extremities. Participants respond to questions on a 1-5 scale (minimum = 8, maximum = 40). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 0.678571429 (4.172694053) | 1.333333333 (5.280630405) | -0.48 (5.393823628)

20. Secondary Outcome: Change From Preoperative Baseline in the Neuro-QOL Item Bank v1.0 "Upper Extremity Function (Fine Motor, ADL)" Short Form
Description: The Neuro-QOL Item Bank v1.0 "Upper Extremity Function (Fine Motor, ADL)" short form evaluates functioning of one's upper extremity function in fine motor and ADL capabilities. Participants respond to questions on a 1-5 scale (minimum = 9, maximum = 45). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 2.392857143 (5.573344536) | 3.896551724 (6.635105918) | 1.76 (5.532329226)

21. Secondary Outcome: Change From Preoperative Baseline in the Neuro-QOL Item Bank v1.0 "Stigma" Short Form
Description: The Neuro-QOL Item Bank v1.0 "Stigma" short form evaluates one's sensitivity of illness-related stigma. Participants respond to questions on a 1-5 scale (minimum = 8, maximum = 40). Higher scores indicate worse function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -2.107142857 (4.755809591) | -2.333333333 (6.143869012) | -1.76 (6.022734706)

22. Secondary Outcome: Change From Preoperative Baseline in the Neuro-QOL Scale v1.0 "Communication" Short Form
Description: The Neuro-QOL Scale v1.0 "Communication" short form evaluates one's difficulty with communication. Participants respond to questions on a 1-5 scale (minimum = 5, maximum = 25). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 0.535714286 (12.79028029) | 1.633333333 (10.9559725) | 2.6 (14.29743567)

23. Secondary Outcome: Change From Preoperative Baseline in the Neuro-QOL Item Bank v1.0 "Emotional and Behavioral Dyscontrol" Short Form
Description: Neuro-QOL Item Bank v1.0 "Emotional and Behavioral Dyscontrol" short form evaluates one's confidence to manage/control symptoms of frustration, disappointment, anger, and other negative emotions. Participants respond to questions on a 1-5 scale (minimum = 8, maximum = 40). Higher scores indicate worse function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -1.142857143 (7.158079019) | 0.133333333 (5.667410364) | -0.76 (7.44020609)

24. Secondary Outcome: Change From Preoperative Baseline in Patient-Reported Outcomes Measurement Information System PROMIS v1.0 "Global Health" Short Form
Description: The PROMIS v1.0 "Global Health" short form evaluates the individual's global health. This is a 10 question scale on which 9 of the questions are answered with a 1 - 5 score. The remaining item is answered with a 0 - 10 score. (minimum = 9, maximum = 55). Higher scores indicate worse function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 1.5 (5.763872155) | 0.433333333 (4.546186984) | 0.375 (4.604463808)

25. Secondary Outcome: Change From Preoperative Baseline in the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.2 "Global Health Mental Health Score"
Description: The (PROMIS) Scale v1.2 "Global Health" evaluates one's overall physical and mental health. This is a 10 item scale with scores ranging from 4-20. Higher scores indicate better overall health.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 2.607142857 (5.983553297) | -0.5 (6.730015115) | 3.166666667 (7.590993901)

26. Secondary Outcome: Change From Preoperative Baseline in Patient-Reported Outcomes Measurement Information System PROMIS v2.0 "Ability to Participate in Social Roles and Activities" Short Form
Description: The PROMIS v2.0 "Ability to Participate in Social Roles and Activities" short form evaluates one's perceived ability to perform one's usual social roles and activities. This is an 8 question measure and answers are given on a 1 - 5 scale (minimum = 8, maximum = 40). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 1.230769231 (5.666093485) | 1.24137931 (5.717486788) | 2.333333333 (5.121707143)

27. Secondary Outcome: Change From Preoperative Baseline in Patient-Reported Outcomes Measurement Information System PROMIS v1.0 "Emotional Distress - Anxiety" Short Form
Description: The PROMIS v1.0 "Emotional Distress - Anxiety" short form evaluates one's feelings of anxiety, such as fear and worry. This is a 7 item scale and participants answer with a 1 - 5 score for each item (minimum = 7, maximum = 35). Higher scores indicate worse function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -2.178571429 (5.192969403) | -0.7 (5.802199345) | -2.333333333 (6.598199139)

28. Secondary Outcome: Change From Preoperative Baseline in Patient-Reported Outcomes Measurement Information System PROMIS v1.0 "Emotional Distress - Depression" Short Form
Description: The PROMIS v1.0 "Emotional Distress - Depression" short form evaluates one's feelings of negative mood and depression. This is an 8 item scale and participants answer with a 1 - 5 score for each item (minimum = 8, maximum = 40). Higher scores indicate worse function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -1.071428571 (4.126953602) | -0.533333333 (4.987801211) | -1.541666667 (7.052468989)

29. Secondary Outcome: Change From Preoperative Baseline in Patient-Reported Outcomes Measurement Information System PROMIS v1.0 "Fatigue" Short Form
Description: The PROMIS v1.0 "Fatigue" short form evaluates one's range of symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. This is a 6 item scale and participants answer with a 1 - 5 score for each item (minimum = 6, maximum = 30). Higher scores indicate worse function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -3.25 (6.304760106) | -1.933333333 (6.766720457) | -2.173913043 (7.088096128)

30. Secondary Outcome: Change From Preoperative Baseline in Patient-Reported Outcomes Measurement Information System PROMIS v2.0 "Physical Function" Short Form
Description: The PROMIS v2.0 "Physical Function" short form measures self-reported capability rather than actual performance of physical activities. This is a 10 item scale and participants answer with a 1 - 5 score for each item (minimum = 10, maximum = 50). Higher scores indicate worse function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 1.964285714 (3.666486287) | 1.724137931 (3.99013562) | 0.652173913 (3.926699929)

31. Secondary Outcome: Change From Preoperative Baseline in Patient-Reported Outcomes Measurement
Description: The PROMIS v1.0 "Pain Interference" short form evaluates the consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. This is a 6 item scale and participants answer with a 1 - 5 score for each item (minimum = 6, maximum = 30). Higher scores indicate worse function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -1.75 (6.304760106) | -2.275862069 (7.372228543) | -2.818181818 (7.768289409)

32. Secondary Outcome: Change From Preoperative Baseline in Patient-Reported Outcomes Measurement Information System PROMIS v1.0 "Sleep Disturbance" Short Form
Description: The PROMIS v1.0 "Sleep Disturbance" short form evaluates one's perceptions of sleep quality. This is an 8 item scale and participants answer with a 1 - 5 score for each item (minimum = 8, maximum = 40). Higher scores indicate worse function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -2.592592593 (7.781928075) | -3.965517241 (8.042222324) | -3.739130435 (4.673108672)

33. Secondary Outcome: Change From Preoperative Baseline in NIH Toolbox Cognition Battery Dimensional Change Card Sort Score
Description: The NIH Toolbox Cognition Battery evaluates cognitive function with Dimensional Change Card Sort Test, Flanker Inhibitory Control and Attention Test, List Sorting Working Memory Test, Picture Vocabulary Test, Pattern Comparison Processing Speed Test, Picture Sequence Memory Test, and Oral Reading Recognition. On this test participants are asked to match pictures to a category and receive one point for each correct match (minimum = 0, maximum = 40). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | 0.210526316 (14.11688881) | 0.473684211 (7.47862451) | 3 (7.874007874)

34. Secondary Outcome: Change From Preoperative Baseline in NIH Toolbox Cognition Battery Flanker Test Score
Description: The NIH Toolbox Cognition Battery evaluates cognitive function with Dimensional Change Card Sort Test, Flanker Inhibitory Control and Attention Test, List Sorting Working Memory Test, Picture Vocabulary Test, Pattern Comparison Processing Speed Test, Picture Sequence Memory Test, and Oral Reading Recognition. The Flanker Test is a test in which participants are asked to focus on a particular stimulus while inhibiting attention to another. An accuracy score is derived by calculating (Accuracy Score = 0.125 * Number of Correct Responses) (minimum=0, maximum=5). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: accuracy score
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
accuracy score | 2.263157895 (8.15026997) | 3.526315789 (4.562752837) | 2.3125 (5.134442521)

35. Secondary Outcome: Change From Preoperative Baseline in NIH Toolbox Cognition Battery List Sorting Working Memory Test Score
Description: The NIH Toolbox Cognition Battery evaluates cognitive function with Dimensional Change Card Sort Test, Flanker Inhibitory Control and Attention Test, List Sorting Working Memory Test, Picture Vocabulary Test, Pattern Comparison Processing Speed Test, Picture Sequence Memory Test, and Oral Reading Recognition. The list sorting working memory test is a test in which lists of items are presented and participants are asked to recall items from the list in a particular order. Scoring is done based on the number of items correctly recalled and sequenced (minimum = 0, maximum = 26). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: change from baseline units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
change from baseline units on a scale | -0.947368421 (9.553787406) | 0.526315789 (11.15232124) | -1.3125 (10.2613758)

36. Secondary Outcome: Change From Preoperative Baseline in NIH Toolbox Cognition Battery Oral Reading Test Score
Description: The NIH Toolbox Cognition Battery evaluates cognitive function with Dimensional Change Card Sort Test, Flanker Inhibitory Control and Attention Test, List Sorting Working Memory Test, Picture Vocabulary Test, Pattern Comparison Processing Speed Test, Picture Sequence Memory Test, and Oral Reading Recognition. The oral reading recognition test is a test in which participants are asked to read and pronounce words as accurately as possible. Pronunciation is judged by the test administrator and a score is given to each response (minimum = 0, maximum = 25). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: words/letters correctly pronounced
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
words/letters correctly pronounced | -1.578947368 (6.890539323) | -1.894736842 (5.867942445) | -3.25 (5.272570531)

37. Secondary Outcome: Change From Preoperative Baseline in NIH Toolbox Cognition Battery Pattern Comparison Test Score
Description: The NIH Toolbox Cognition Battery evaluates cognitive function with Dimensional Change Card Sort Test, Flanker Inhibitory Control and Attention Test, List Sorting Working Memory Test, Picture Vocabulary Test, Pattern Comparison Processing Speed Test, Picture Sequence Memory Test, and Oral Reading Recognition. The pattern comparison test is a test in which participants are presented with two pictures and are asked to discern whether they are he same or different. Correct answers are given one point for up to a maximum of 130 trials (minimum = 0, maximum = 130). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
units on a scale | 1.421052632 (11.19680406) | 3.526315789 (13.61114095) | 2.8125 (14.27920983)

38. Secondary Outcome: Change From Preoperative Baseline in NIH Toolbox Cognition Battery Picture Sequencing Test Score
Description: The picture sequencing test is a test of episodic memory in which participants are asked to recall increasingly lengthy series of illustrated objects and activities that are presented in a particular order on a computer screen. Participants are given credit for each adjacent pair of pictures they correctly place up to the maximum value for the sequence, which is one less than the sequence length (minimum = 0, maximum = 105). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: number of correct sequences identified
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
number of correct sequences identified | 1.842105263 (13.22146049) | 4.263157895 (10.09863635) | 2.875 (8.891006692)

39. Secondary Outcome: Change From Preoperative Baseline in NIH Toolbox Cognition Battery Picture Vocabulary Test Score
Description: The NIH Toolbox Cognition Battery evaluates cognitive function with Dimensional Change Card Sort Test, Flanker Inhibitory Control and Attention Test, List Sorting Working Memory Test, Picture Vocabulary Test, Pattern Comparison Processing Speed Test, Picture Sequence Memory Test, and Oral Reading Recognition. The picture vocabulary test is a test in which participants are presented with an audio recording of a word and four photographic images on the computer screen and asked to select the picture that most closely matches the meaning of the word (minimum = 0, maximum = 25). Higher scores indicate better function.
  A change between baseline and performance at 2, 4, and 6 months post surgery is reported here. Score calculation is baseline - performance while on directional DBS guided by behavior, baseline - performance while on omnidirectional DBS guided by behavior, and baseline - performance while on directional DBS guided by biomarkers.
Time Frame: 2, 4, and 6 months post op
Population: All participants experienced all three arms of the crossover study.
Measure: Mean (Standard Deviation); unit: number of correct matches
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
Number analyzed (Participants) | 31 | 31 | 31
number of correct matches | -1.105263158 (5.205709866) | -0.578947368 (5.480427695) | -1.0625 (5.93822364)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Directional DBS Guided by Behavior | Omnidirectional DBS Guided by Behavior | Directional DBS Guided by Biomarkers
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 3/31 | 4/31 | 0/31
Other Adverse Events (participants affected / at risk) | 2/31 | 0/31 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Directional DBS Guided by Behavior (N=31) | Omnidirectional DBS Guided by Behavior (N=31) | Directional DBS Guided by Biomarkers (N=31)
SAE1 (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Myocardial infarction
SAE2 (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) — DBS lead placed suboptimally
SAE3 (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Postoperative seizure
SAE4 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Panic attack
SAE5 (Product Issues) | 1 (1) | 1 (1) | 0 (0) — Separation of product components post surgery
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Directional DBS Guided by Behavior (N=31) | Omnidirectional DBS Guided by Behavior (N=31) | Directional DBS Guided by Biomarkers (N=31)
AE1 (Product Issues) | 2 (2) | 0 (0) | 0 (0) — Short circuit between DBS contacts

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT03353688/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03353688/SAP_002.pdf